CLINICAL TRIAL: NCT00645294
Title: A Phase 1-2 Open-Label Study of the Pharmacokinetics and Safety of a Single Dose of Adefovir Dipivoxil in Children and Adolescents (Aged 2-17) With Chronic Hepatitis B
Brief Title: Open Label Study of Pharmacokinetics and Safety of Dose of Adefovir Dipivoxil in Children and Adolescents With HBV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Elsa Mondou, MD, Gilead Sciences
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GS-02-517
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Adefovir dipivoxil; Children; Adolescents; Pharmacokinetics
MeSH Terms: conditions — Hepatitis B | interventions — adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Group A (Other): ADV (0.14 mg/kg) oral suspension formulation on Day 1 followed by ADV (0.3 mg/kg) oral suspension formulation on Day 8 in 2-6 and 7-11 year old age group
  Interventions: Drug: Adefovir dipivoxil
- Treatment Group B (Other): ADV (0.3 mg/kg) oral suspension formulation on Day 1 followed by ADV (0.14 mg/kg) oral suspension formulation on Day 8 in 2-6 and 7-11 year old age group
  Interventions: Drug: Adefovir Dipivoxil
- Treatment Group C (Other): ADV 10 mg single dose on Day 1 in 12-17 year old age group
  Interventions: Drug: Adefovir Dipivoxil

INTERVENTIONS:
Drug: Adefovir dipivoxil — 0.14 mg/kg on Day 1, followed by 0.3 mg/kg on Day 8
  Arms: Treatment Group A
Drug: Adefovir Dipivoxil — 0.3 mg/kg on Day 1, followed by 0.14 mg/kg on Day 8
  Arms: Treatment Group B
Drug: Adefovir Dipivoxil — ADV 10 mg on Day 1
  Arms: Treatment Group C

SUMMARY:
Open-label study of the pharmacokinetics of adefovir dipivoxil in children and adolescents infected with chronic hepatitis B.

DETAILED DESCRIPTION:
Children and adolescents with chronic hepatitis B and compensated liver, HBeAg-positive and serum HBV DNA positive (greater than or equal to 1 x 100,000 copies/mL by Roche Amplicor Monitor PCR) received doses of adefovir dipivoxil in a cross-over design. Subjects aged 2-11 received two single doses (0.14 mg/kg and 0.3 mg/kg liquid formulation) and subjects 2-17 received one dose (10 mg liquid formulation).

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 2 and 17 (inclusive) with chronic hepatitis B as evidenced by the following:
* HBsAg positive for a minimum of 6 months
* HBeAg positive and HBV DNA greater than or equal to 1 x 100,000 copies/mL at screening
* Children and adolescents with compensated liver disease
* ALT levels greater than or equal to 1.2 upper limit of normal (applicable to 7- to 17-year-old children and adolescents only)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2003-02; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
To characterize the PK profile of adefovir 0.14 mg/kg and 0.3 mg/kg in children 2-11 years, including dose proportionality of adefovir dipivoxil liquid formulation. To characterize the PK profile of adefovir dipivoxil 10 mg in adoloscents 12-17 years. | 8 days

CONTACTS AND LOCATIONS:
Locations (10):
- Cliniques Universitaries, Brussels, Belgium
- Germany (5):
  - J.W. Goethe-Universitat, Frankfurt
  - Mid. Hochschule Hannover Kinderklinik, Hanover
  - Kinderklinik der Gutenberg Universitat, Mainz
  - Standort Lindwurmstrasse, München
  - Zentrum fur Kinder und Jugendmedizin der Klinikum, Wuppertal
- Poland (2):
  - Oddzial Chorob Infekcyjnych Dzieci, Krakow
  - Klinika Gastroenterologii, Warsaw
- United Kingdom (2):
  - King's College Hospital, London, England
  - University of Birmingham, Birmingham